CLINICAL TRIAL: NCT02191449
Title: Influence of Warfarin on Thromboelastography and Transfusion
Brief Title: The Influence of Preoperative Warfarin Medication on Thromboelastography and Blood Transfusion
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: KUH1160068
Record Dates: First submitted 2014-06-29; First posted 2014-07-16 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Warfarin therapy is usually monitored using the international normalized ratio (INR), and prolonged INR means coagulation impairment that can leads elevating transfusion requirement after operation. This study was designed to assess the relationships with warfarin and TEG values related to transfusion amount, to set up blood transfusion strategy in patients on atrial fibrillation undergoing cardiac surgery.

DETAILED DESCRIPTION:
This study was a retrospective evaluation of patients who have received cardiac surgery with Maze-operation from March 2008 to November 2013.

Patients who have atrial fibrillation undergoing cardiac surgery with Maze-operation were included.

The following exclusion criteria are applied:

1. Patients who have taken medicine related to coagulation (such as antiplatelets like aspirin and clopidogrel) except warfarin or bridged heparin
2. Patients whose laboratory values could not be confirmed by medical records review.

Patients were categorized by two groups.

1. W group: patients on atrial fibrillation who have taken warfarin for p.o medication.
2. C group: patients on atrial fibrillation who have not taken warfarin for p.o medication.

Using blood sample, authors examined as follows:

1. Preoperative (maximum 5days before operation) and postoperative (30min after ICU admission) coagulation values with haematologic values: PT/aPTT, INR, Hb, Hct, platelet levels.
2. ROTEM values at 30min after anaesthetic induction and 30min after ICU admission: Clotting time (CT), clot formation time (CFT), maximum clot firmness (MCF), maximum lysis (ML)
3. Intraoperative (during operation) and postoperative (during admission, an expected average of 5 weeks) total transfusion amount: RBC, FFP, PC, cryoprecipitate.
4. Post operative 24 hr bleeding amount in the chest tube drain bottle.
5. The duration (maximum 2 weeks) of warfarin discontinuation. (in W group)

Statistical analysis was performed using unpaired t-test and chi-square test to compare patients demographic data and other parameters. To determine the relationship of INR and ROTEM parameters with bleeding amount and transfusion amount, multiple linear regression model that accounted for all confounder variables was used. For each factor in the multiple regression model, variables with a p value of less than 0.10 were kept in the final model. The data was analyzed using the program Statistical Package for the Social Sciences ver. 18.0 (SPSS Inc, Chicago, USA). A value of p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have atrial fibrillation undergoing cardiac surgery with Maze-operation.

* W group : Patients who have had warfarin therapy before operation due to treat Atrial fibrillation
* C group : Patients who have not had warfarin therapy before operation

Exclusion Criteria:

* 1. Patients who have taken medicine related to coagulation (such as antiplatelets like aspirin and clopidogrel) except warfarin or bridged heparin.
* 2. Patients whose laboratory values could not be confirmed by medical records review.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery with Maze-operation
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Rotational Thromboelastography : Clotting time (CT) | 30min after anesthetic induction and 15 mins after CPB weaning status

SECONDARY OUTCOMES:
Rotational Thromboelastography : clot formation time (CFT) | 30min after anesthetic induction and 15 mins after CPB weaning status

OTHER OUTCOMES:
Rotational Thromboelastography : maximum clot firmness (MCF) | 30min after anesthetic induction and 15 mins after CPB weaning status
Rotational Thromboelastography : maximum lysis (ML) level Rotational Thromboelastography : maximum lysis (ML) level | 30min after anesthetic induction and 15 mins after CPB weaning status
amount of Blood transfusion | intraoperative (during operation) and postoperative (during admission, an expected average of 5 weeks)
Coagulation values : preprothrombin time (PT) | preoperative (maximum 5days before operation) and postoperative (30min after ICU admission)
Coagulation values : activated partial thromboplastin time (aPTT) | preoperative (maximum 5days before operation) and postoperative (30min after ICU admission)

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D,Ph.D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea